CLINICAL TRIAL: NCT00565552
Title: Influence of a Silicone Gel (Dermatix®) on Thoracic Scar Formation After Harvesting of Autologous Rib Cartilage for Standardised Total Ear Reconstruction
Brief Title: Influence of a Silicone Gel (Dermatix®) on Thoracic Scar Formation After Harvesting of Autologous Rib Cartilage
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Schleswig-Holstein (Other)
Responsible Party: Dr. Stefan Nitsch, University of Schleswig-Holstein
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Dermatix01
Record Dates: First submitted 2007-11-29; First posted 2007-11-30 (Estimated); Last update posted 2007-11-30 (Estimated); Status verified 2007-11

CONDITIONS: Cicatrix, Hypertrophic; Keloid
Keywords: silicone gel; cicatrix; wound healing; scar; keloid
MeSH Terms: conditions — Cicatrix, Hypertrophic; Keloid; Cicatrix | interventions — Silicone Gels

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Active Comparator): Each patient uses the silicone gel on one half of the scar, leaving the other one blank as an internal control.
  Interventions: Drug: Silicone gel (Dermatix®)

INTERVENTIONS:
Drug: Silicone gel (Dermatix®) — The half one the scar to treat was randomised among patients. After regular cleaning of the skin around the scar one half was thinly creamed with the silicone gel from medial to lateral and let dry for 5 minutes. It was done twice daily.
  Other Names: Dermatix®

SUMMARY:
So far the evaluation of scar treatment was based on subjective criteria. The patient groups were divided into treated versus non-treated.

In this study we use patients undergoing ear reconstruction with autologous rib cartilage. The thoracic scar of harvesting the rib cartilage is routinely reopened after 3 month during second stage of reconstruction. Therefore we have a ideal model of clinical, physiological and histological scar evaluation in a homologous patient group.

All patients randomly treat one half of the scar with a silicone gel (Dermatix). The other half is untreated as an internal control.

ELIGIBILITY:
Inclusion Criteria:

* patients with high grade microtia requiring a reconstruction with autologous rib cartilage

Exclusion Criteria:

* diabetes mellitus
* vascular disease
* known allergic reaction to silicone

Min Age: 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2007-01; Study Completion 2009-01 (Estimated)

PRIMARY OUTCOMES:
Beausang's scar scale, skin elasticity (Cutometer®), skin moisture (Corneometer®), skin color (Chromameter®, Mexameter®), histological evaluation (HE, elastica, actin etc.) | 45 minutes

SECONDARY OUTCOMES:
allergic reaction compliance | retrospective

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Nitsch, MD, Principal Investigator — University Hospital Schleswig-Holstein
Locations (1):
- University Hospital Schleswig-Holstein, Lübeck, Germany